CLINICAL TRIAL: NCT06027983
Title: Phase IB Followed by Phase II Study of Trastuzumab Combined With Autologous Chimeric Receptor T Cells in HER2+ Advanced Breast Cancer and Other Solid Tumors
Brief Title: Chimeric Receptor T Cells With Trastuzumab in HER2+ Advanced Breast Cancer and Other Solid Tumors
Status: Not yet recruiting | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National University Hospital, Singapore (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: ACEHER2
Record Dates: First submitted 2023-08-31; First posted 2023-09-07 (Actual); Last update posted 2025-09-23 (Actual); Status verified 2025-08

CONDITIONS: HER2+ Advanced Breast Cancer; Other Solid Tumors
MeSH Terms: interventions — Trastuzumab; fludarabine

STUDY DESIGN:
Intervention Model Description: This is a single arm, open-label, phase Ib safety lead in, followed by phase II study. The phase Ib segment will be carried out in a standard 3+3 dose escalation design. In the phase II, dose expansion will be carried out to a total of 10 patients at recommended phase II dose in both phase Ib and II.
  Phase Ib: Patients with advanced solid tumors will be enrolled in a 3+3 dose escalation fashion, with projected enrolment of between 6-30 patients to determine RP2D. Once the RP2D is confirmed, the study will proceed to phase II.
  Phase II: Up to a total of 10 patients with HER2+ advanced breast cancer will be enrolled.
  For patients who are in Dose level 3 - 5 will require additional Trastuzumab,erythropoietin beta and Lymphodepletion.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (1):
- Chimeric Receptor T-cells (Experimental): Eligible patients will undergo apheresis prior to cycle 1 therapy. Treatment comprises of trastuzumab followed by chimeric receptor T-cells in cycle 1.
  During Cycle 2 onwards till disease progression, patients will receive IV or SC trastuzumab only, every 3 weeks.
  Interventions: Drug: Chimeric receptor T-cells + Trastuzumab; Drug: Fludarabine and Cyclophosphosphamide

INTERVENTIONS:
Drug: Chimeric receptor T-cells + Trastuzumab — Chimeric receptor T-cells will be administered by infusion. Trastuzumab will be administered intravenously.
Drug: Fludarabine and Cyclophosphosphamide — 3-day chemotherapy regimen of fludarabine and cyclophosphamide for lymphodepletion
  Other Names: Lymphodepletion

SUMMARY:
This phase Ib study aims to assess the safety and feasibility of combination of chimeric receptor T cells with trastuzumab in patients with HER2+ solid tumors, with further expansion of study population in HER2+ metastatic breast cancer once safety has been established.

DETAILED DESCRIPTION:
Hypothesis

Investigators hypothesize that trastuzumab-mediated cytotoxicity will be augmented by the infusion of autologous chimeric receptor T-cells.

Primary Objectives

1. To determine the safety of autologous chimeric receptor T-cells in patients with HER2+ advanced solid tumors
2. To determine the clinical benefit rate (CBR) of autologous chimeric receptor T-cells in patients with HER2+ advanced breast cancer

Secondary Objectives

1. To determine the expansion and persistence of autologous chimeric receptor T-cells after a single infusion in patients with advanced solid tumors
2. To determine anti-tumor efficacy in terms of objective response rate (ORR) and progression-free survival (PFS) of autologous chimeric receptor T-cells in patients with HER2+ advanced breast cancer

ELIGIBILITY:
Inclusion Criteria:

Patients may be included in the study only if they meet all of the following criteria:

* Age ≥ 21 years.
* Histologically confirmed diagnosis of HER2-positive cancer defined by immunohistochemistry (IHC) to be HER2 IHC3+ or HER2 IHC2+ and FISH positive. If immunohistochemistry is not available, FISH method is acceptable. The HER2 positivities by FISH is determined as FISH amplification ratio positive by institutional guidelines. Tumor subtype for each phase include :
* Phase I: HER2-positive breast or gastric cancer or other treatment-refractory HER2-positive solid tumors
* Phase II : HER2-positive breast carcinoma
* Eastern Cooperative Oncology Group (ECOG) performance status 0-1.
* Has measurable or evaluable disease based on RECIST 1.1 criteria
* Estimated life expectancy of at least 12 weeks.
* Prior lines of therapy:
* HER2-positive breast cancer - patient must have failed at least two lines of anti-HER2 based therapy for advanced/metastatic cancer. Patients with documented relapse while receiving or within 6 months of completion of adjuvant or neoadjuvant trastuzumab for HER2-positive breast cancer will be considered as 1 prior line of therapy.
* HER2-positive gastric cancer - patient must have failed at least one line of anti-HER2 based therapy.
* Other refractory HER2-positive solid tumors (non-breast, non-gastric) - have no standard therapies or have failed or unable to tolerate standard therapies
* Has recovered from acute toxicities from prior anti-cancer therapies
* Left ventricular ejection fraction ≥50%
* Adequate organ function including the following:

  o Bone marrow: Absolute neutrophil (segmented and bands) count (ANC) ≥ 1.5 x 109/L Platelets ≥ 100 x 109/L Haemoglobin ≥ 8 x 109/L

  o Hepatic: Bilirubin ≤ 1.5 x upper limit of normal (ULN), ALT or AST≤ 2.5x ULN, (or ≤5 X with liver metastases)

  o Renal: Creatinine ≤ 1.5x ULN
* Signed informed consent from patient or legal representative.
* Able to comply with study-related procedures.
* Specific to cohorts 3, 4 and 5 : Patients who have a history of VTE are eligible if as long as they are receiving therapeutic/prophylactic doses of anticoagulation.

Exclusion Criteria:

Patients will be excluded from the study for any of the following reasons:

* Treatment within the last 30 days with any investigational drug.
* Concurrent administration of any other tumour therapy, including cytotoxic chemotherapy, hormonal therapy, and immunotherapy.
* Major surgery within 28 days of study drug administration.
* Active infection that in the opinion of the investigator would compromise the patient's ability to tolerate therapy.
* Pregnancy.
* Breast feeding.
* Serious concomitant disorders that would compromise the safety of the patient or compromise the patient's ability to complete the study, at the discretion of the investigator.
* Active bleeding disorder or bleeding site.
* Non-healing wound.
* Poorly controlled diabetes mellitus.
* Second primary malignancy that is clinically detectable at the time of consideration for study enrolment.
* Symptomatic brain metastasis.
* History of significant neurological or mental disorder, including seizures or dementia,
* History of autoimmune disease or use of gamma immunoglobulin
* Unable to comply with study procedures

Ages: 21 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 36 (Estimated)
Dates: Start 2026-11-01 (Estimated); Primary Completion 2026-12-31 (Estimated); Study Completion 2027-12-31 (Estimated)

PRIMARY OUTCOMES:
Time to treatment failure | 3 years
  defined as the time from the date of study enrolment to the date of the first of the following events: early discontinuation of study therapy, progressive disease, or death due to any cause. Time to treatment failure will be censored at the date of the last follow-up visit for patients who did not discontinue early, who are still alive, and who have not progressed.
Progression-free survival | 3 Years
  is defined as the time from the date of study enrolment to the first date of documented disease progression. Progression-free survival will be censored at the date of death for patients who have not had documented disease progression. For patients who are still alive at the time of analysis and who have not had documented disease progression, progression-free survival will be censored at the date of the last follow-up visit.
Duration of tumour response | 3 Years
  Among tumor responders, the duration of tumor response is measured from the date of enrolment until the first date of documented disease progression or death due to any cause, whichever occurs first. Duration of tumor response will be censored at the date of the last follow-up visit for tumor responders who are still alive and who have not progressed.

CONTACTS AND LOCATIONS:
Overall Officials: Soo Chin Lee, Principal Investigator — National University Hospital, Singapore

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Lee SC, Shimasaki N, Lim JSJ, Wong A, Yadav K, Yong WP, Tan LK, Koh LP, Poon MLM, Tan SH, Ow SGW, Bharwani L, Yap YS, Foo MZQ, Coustan-Smith E, Sundar R, Tan HL, Chong WQ, Kumarakulasinghe NB, Lieow JLM, Koe PJX, Goh BC, Campana D. Phase I Trial of Expanded, Activated Autologous NK-cell Infusions with Trastuzumab in Patients with HER2-positive Cancers. Clin Cancer Res. 2020 Sep 1;26(17):4494-4502. doi: 10.1158/1078-0432.CCR-20-0768. Epub 2020 Jun 10. PMID 32522887